CLINICAL TRIAL: NCT04834206
Title: Induction Chemotherapy With Nedaplatin, Docetaxel and 5-Fluorouracil Followed by Concurrent Nedaplatin and Radiotherapy in Locoregionally Advanced Nasopharyngeal Carcinoma: a Single Arm, Open Label, Multicenter, Phase II Clinical Study.
Brief Title: Nedaplatin in Treatment for Nasopharyngeal Carcinoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Affiliated Cancer Hospital & Institute of Guangzhou Medical University (Other)
Responsible Party: Principal Investigator, Jin-Quan Liu, Section Chief, Affiliated Cancer Hospital & Institute of Guangzhou Medical University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NPC-NDP-SGL arm
Record Dates: First submitted 2021-04-01; First posted 2021-04-08 (Actual); Last update posted 2022-05-10 (Actual); Status verified 2022-05

CONDITIONS: Nasopharyngeal Carcinoma
Keywords: Induction chemotherapy; Nedaplatin; Concurrent chemoradiotherapy; Nasopharyngeal Carcinoma
MeSH Terms: conditions — Nasopharyngeal Carcinoma | interventions — Docetaxel; nedaplatin; Fluorouracil

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- DNF-N (Other): 1. Induction chemotherapy:
     three cycles of intravenous docetaxel 60 mg/m² on day 1, intravenous nedaplatin 60 mg/m² on day 1, and continuous intravenous fluorouracil 600 mg/m² per day from day 1 to day 5, every 3 weeks
  2. Concurrent chemoradiotherapy:
     three cycles of 100 mg/m² nedaplatin every 3 weeks, concurrently with intensity-modulated radiotherapy
  3. Radiotherapy: radical intense modulated radiation therapy
  Interventions: Drug: Docetaxel, nedaplatin, fluorouracil; Radiation: IMRT; Drug: Nedaplatin

INTERVENTIONS:
Drug: Docetaxel, nedaplatin, fluorouracil — Induction chemotherapy. Docetaxel 60 mg/m2 intravenous day1. Nedaplatin 60 mg/m2 intravenous day1. Fluorouracil 3000 mg/m2 continuous intravenous infusion 120 hours from day1. Every 21 days, 3 cycles.
  Other Names: DNF
Radiation: IMRT — Intensity modulated-radiotherapy (IMRT) is given as 2.0-2.33 Gy per fraction with five daily fractions per week for 6-7 weeks to a total dose of 66 Gy or greater to the primary tumor.
  Other Names: RT
Drug: Nedaplatin — Concurrent chemotherapy. nedaplatin 100 mg/m2 intravenous at day1, 22, 43 of radiotherapy.
  Other Names: N

SUMMARY:
To evaluate the efficacy of induction chemotherapy with nedaplatin, docetaxel and 5-Fluorouracil followed by concurrent nedaplatin combined with radical radiotherapy in locally advanced nasopharyngeal carcinoma.

DETAILED DESCRIPTION:
This is a prospective, phase II clinical trial to evaluate the efficacy and safety of induction chemotherapy with nedaplatin, docetaxel and 5-Fluorouracil followed by concurrent nedaplatin combined with radical radiotherapy in locally advanced nasopharyngeal carcinoma patients. This is a multicenter study. All patients will be enrolled in endemic area. All patients will receive radical intense modulate radiation therapy (IMRT). The primary endpoint is objective response rate (ORR).

ELIGIBILITY:
Inclusion Criteria:

* Patients with newly histologically confirmed non-keratinizing nasopharyngeal carcinoma, including WHO II or III
* Original clinical staged as III-IVa (except T3-4N0) according to the 8th edition American Joint Committee on Cancer staging system
* No evidence of distant metastasis (M0)
* Age between 18-65
* WBC≥4×10^9/ l, platelet ≥ 100×10^9/ l and hemoglobin ≥ 90g/l
* With normal liver function test (TBIL、ALT、AST ≤ 2.5×uln)
* With normal renal function test (creatinine ≤ 1.5×uln or ccr ≥ 60ml/min)
* Satisfactory performance status: KARNOFSKY scale (KPS) > 70
* Patients must give signed informed consent

Exclusion Criteria:

* Treatment with palliative intent
* The primary tumor or lymph node has undergone chemotherapy or surgery (except operations for diagnostic purposes)
* Prior malignancy except adequately treated basal cell or squamous cell skin cancer, in situ cervical cancer
* History of previous radiotherapy, chemotherapy, or surgery (except diagnostic) to the primary tumor or nodes
* History of previous radiotherapy
* Pregnancy or lactation
* Any severe intercurrent disease, which may bring unacceptable risk or affect the compliance of the trial, for example, unstable cardiac disease requiring treatment, acute exacerbation of chronic obstructive pulmonary disease or other respiratory illness requiring admission to hospital, active hepatitis, and mental disturbance.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2021-05-01 (Actual); Primary Completion 2021-10-29 (Actual); Study Completion 2022-05-01 (Actual)

PRIMARY OUTCOMES:
objective response rate (ORR) | at the end of radiotherapy(±1week）
  CR+PR

SECONDARY OUTCOMES:
Overall Survival(OS) | 3 years
  The OS was defined as the duration from the date of beginning of treatment to the date of death from any cause or censored at the date of the last follow-up.
Progress-Free Survival (PFS) | 3 years
  Progress-free survival is calculated from the date of beginning of treatment to the date of locoregional failure, distant failure, or death from any cause, whichever occurred first.
Locoregional Relapse-Free Survival(LRRFS) | 3 years
  Relapse-free survival was defined as the time from beginning of treatment to local or regional relapse, or death from any cause.
Distant metastasis-Free Survival(DMFS) | 3 years
  Distant metastasis-free survival was defined as the time from beginning of treatment to distant metastasis, or death from any cause.
Quality of life (QoL) | 3 years
  Quality of life (QoL) was assessed using the European Organization for Research and Treatment of Cancer Quality of Life Questionnaire module for head and neck (EORTC QLQ-H&N35). The EORTC QLQ-H&N35 scale employs a 4-point response format ("not at all" to "very much"). Scale scores are transformed to a scale from 0 to 100 according to the EORTC scoring algorithm. For the functioning and the global QoL scale, a higher score indicates better health. For the symptom scales, a higher score indicates a higher level of symptom burden. Either English or Chinese version will be used according to patient's language habits.

CONTACTS AND LOCATIONS:
Overall Officials: Jinquan Liu, M.D, Study Director — Affiliated Cancer Hospital & Institute of Guangzhou Medical University
Locations (1):
- Department of radiotherapy(Section 5),Affiliated Cancer Hospital & Institute of Guangzhou Medical Universityedical University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Chen FZ, Deng Y, Yin WJ, Wang MY, Yang F, Yang ZH, Zhou LP, Chen SD, Chen JL, Jiang XZ, Zhou AX, Ou YM, Liu JQ, Chen DP, Qi B. Induction chemotherapy with nedaplatin, docetaxel and 5-fluorouracil followed by concurrent nedaplatin and radiotherapy in locoregionally advanced nasopharyngeal carcinoma: A single arm, open label, phase II clinical trial. Transl Oncol. 2026 Feb;64:102634. doi: 10.1016/j.tranon.2025.102634. Epub 2026 Jan 6. PMID 41496409